CLINICAL TRIAL: NCT00586235
Title: Registration and Fusion of Real-Time Ultrasound With CT for Lesion Localization and Characterization
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Siemens Medical Solutions (Industry)
Responsible Party: Principal Investigator, Matthew R. Callstrom, Study Prinicple Investigator, Mayo Clinic
Other Study IDs: 06-002982; 06-002982
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Kidney or Liver Tumors
Keywords: Fusion; Ultrasound; Computed tomography
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: patients with indeterminate kidney or liver lesions

SUMMARY:
Acquire CT data and US and transducer position data (magnetic sensor system) of focal hepatic or renal lesions to serve as sample data sets for fusion algorithm development and subsequent optimization.

DETAILED DESCRIPTION:
Acquire CT data and US and transducer position data (magnetic sensor system) of focal hepatic or renal lesions to serve as sample data sets for fusion algorithm development and subsequent optimization.

Optimize image fusion algorithms for use in goal. Develop registration algorithms that result in maximal lesional overlap with a clinically relevant difference in an epicenter location of ≤ 2 cm for lesional identification and, ultimately ≤ 0.3 cm for interventional procedures.

ELIGIBILITY:
Inclusion Criteria:

* Focal lesion involving the liver or kidney bases on CT or MRI Imaging
* Liver lesion size >5 mm and <5 cm in diameter or renal lesion size is >5 mm and <4 cm in diameter
* Age >18 years old
* Patient has provided written informed consent

Exclusion Criteria:

* Patient with cardiac pacemaker or defibrillator
* Pregnant or lactating woman
* Patient with severe IV contrast allergy (previous reaction to IV contrast not mitigated by appropriate premedication)
* Patient unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with kidney or liver tumors
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2007-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Primary Endpoints: Global Fiducial Registration Error (FRE) of real-time US and fused CT images, Target Registration Error (TRE) and distance between lesional epicenters of real-time US and fused CT images. | 2 years

SECONDARY OUTCOMES:
Secondary Endpoint: Number of coregistration attempts to realize separation of lesional epicenters of real-time US and fused CT images of ≤2 cm and the number of attempts to realize a separation of ≤0.3 cm. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R. Callstrom, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials